CLINICAL TRIAL: NCT01850771
Title: A Single-Blinded, Randomized Controlled Trial of Regenexx™ PL-Disc Versus Steroid Epidurals for Treatment of Lumbar Radiculopathy
Brief Title: Regenexx™ PL-Disc Versus Steroid Epidurals for Lumbar Radiculopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruitment
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RSI2013-RCT02
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Radiculopathy; Herniated Disc; Disc Degeneration
Keywords: Lumbar Radiculopathy; Disc bulge; Disc herniation; Disc degeneration
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Displacement; Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regenexx PL-Disc (Active Comparator): Injection of Regenexx PL-Disc into the epidural space once a week for two weeks.
  Interventions: Procedure: Regenexx PL-Disc
- Steroid Epidural (Active Comparator): Injection of steroid into the epidural space once a week for two weeks
  Interventions: Procedure: Steroid Epidural

INTERVENTIONS:
Procedure: Regenexx PL-Disc — Injection into the epidural space under image guidance of autologous, concentrated peripheral blood based platelet mix combined with a nanogram dose of corticosteroid.
  Arms: Regenexx PL-Disc
Procedure: Steroid Epidural — Injection into the epidural space under image guidance of 3 mg of betamethasone.
  Arms: Steroid Epidural

SUMMARY:
The primary objective of this study is to compare the improvement in subject-reported clinical outcomes for Regenexx PL-Disc vs. steroid epidural for treatment of lumbar radiculopathy, from baseline to 3 months, with continued evaluation of efficacy and durability up to 12 months.

Secondary objectives include incidence of post-operative complications, adverse events, re-injections, and surgical intervention; change in pain score and use of pain medications.

DETAILED DESCRIPTION:
Prospective, single-blinded, randomized, controlled to include 25 subjects treated with Regenexx PL-Disc and 25 subjects treated with steroid epidural injection with the steroid epidural group crossing over to the PL-Disc injection group at 3 months.

Subjects will have symptoms consistent with lumbar radiculopathy confirmed by physical examination.

Subjects will be enrolled within 60 days prior to injection and take part in follow-up visits for one year following treatment. A preoperative visit will occur at the time of enrollment; follow-up visits will occur at the clinical site at 6 weeks, 3 months, 6 months and 12 months post injection. Subjects will remain blinded to the treatment allocation through at least the 3 month primary endpoint. Control subjects not improving after the 3 month visit will be unblinded and given the opportunity to cross-over to the PL-Disc group.

Subjects will complete the study following the 1 year follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Pain, spasm, or functional disability in the low back and diagnosed as radiculopathy having failed conservative treatment (e.g. NSAIDs, physician initiated physical therapy) for at least 3 months and not longer than 2 years
* Significant functional disability related to pain, lack of strength, or other back or leg symptoms
* Physical examination consistent with lumbar radiculopathy
* Lumbar disc bulge, herniation, and/or Kader grade 2 or greater multifidus atrophy evident on MRI and consistent with physical exam findings
* Is independent, ambulatory, and can comply with all post-operative evaluations and visits

Exclusion Criteria:

* Symptomatic central or foraminal stenosis
* Previous low back surgery
* Prior epidural steroid injection or other low back injection therapy within the past year
* >50% loss of disc height at the symptomatic level
* Spondylolisthesis
* Inflammatory or auto-immune based pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout)
* Quinolone or Statin induced myopathy/tendinopathy
* Severe neurogenic inflammation of the cutaneous nerves
* Condition represents a worker's compensation case
* Currently involved in a health-related litigation procedure
* Is pregnant
* Bleeding disorders
* Currently taking anticoagulant or immunosuppressive medication
* Allergy or intolerance to study medication
* Use of chronic opioid,
* Documented history of drug abuse within six months of treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index Change from Baseline | Change from baseline to 3 months
  The primary endpoint for this study is the difference between treatment groups in the within patient mean change from baseline to 3 months in Oswestry Disability Index (ODI) scores.

SECONDARY OUTCOMES:
Mean Functional Rating Index Scores | 6 weeks, 3 months, 6 months, 12 months
  Difference between treatment groups in mean Functional Rating Index (FRI) scores at each follow-up timepoint.
Mean ODI scores | 6 weeks, 3 months, 6 months, 12 months
  Difference between treatment groups in mean ODI scores at each follow-up timepoint
Mean Pain Scales | 6 weeks, 3 months, 6 months, 12 months
  Difference between treatment groups in mean 0-10 pain scales at each follow-up timepoint
Incidence of Complications and Adverse Events | 12 months
  Incidence of post-operative complications and adverse events between treatment groups.
Incidence of re-injection/re-operation | 12 months
  Incidence of re-injection and surgical operation between treatment groups.
Use of pain medications | 6 weeks, 3 months, 6 months, 12 months
  Difference between treatment groups in use of pain medications at each follow-up timepoint
Time to Resolution of Complications and Adverse Events | 12 months
  Time to resolution of post-operative complications and adverse events between treatment groups.
Time to re-injection/re-operation | 12 months
  Time to re-injection and surgical operation between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Centeno-Schultz Clinic
Locations (1):
- Centeno-Schultz Clinic, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No